CLINICAL TRIAL: NCT05666596
Title: Do Advanced Hybrid Closed Loop Systems Effect Nutrient Intake?: Short Term Follow-up Study, Real Life Data
Brief Title: Do Advanced Hybrid Closed Loop Systems Effect Nutrient Intake?: Real Life Data
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yasemin Atik Altinok, Dietician, PhD, Ege University
Other Study IDs: AHCLS T1D
Record Dates: First submitted 2022-12-02; First posted 2022-12-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This 6-month follow-up study was conducted to investigate the effect of AHCLS on the energy and macronutrient intake of children, adolescents, and young adults with Type 1 diabetes (T1D). All participants with T1D on an AHCLS (MiniMed 780GTM) receiving care at the Pediatric Endocrinology and Diabetes Clinic of Ege University (Izmir, Turkey) were eligible for the study. The children and adolescents with T1D with at least 3 days of food diary available before AHCLS and at 3rd and 6th months at AHCLS were included in the study

DETAILED DESCRIPTION:
In all participants, height was measured to the nearest centimeter using a rigid stadiometer. Weight was measured unclothed to the nearest 0.1 kg using a calibrated balance scale. Body mass index (BMI) was calculated by the weight (kg)/height (m²) equation. Standard deviation scores (SDS) for weight, height, and BMI were calculated according to age and gender using reference values for Turkish children and adolescents (1). For young adults, a BMI of 18.5-24.9 kg/ m² is considered normal weight Participants recorded all food and beverage (including dressings) consumed and the servings reported by weight, before and after (3rd, 6th month) switching to MiniMed 780GTM. Before entering data in the nutrient analysis program, the research team dietician reviewed all completed diet records and asked for supplementary information if needed. The analysis included 1076 snacks and meals (750 meals, 326 snacks) dietary records. Total energy intake (kcal), fat (energy %), protein (energy %), carbohydrate (energy %), saturated fatty acids (energy %), cholesterol (mg), and dietary fiber (g/1000 kcal) intake were calculated using the Ebispro for Windows,; Turkish Version (BeBiS 8.2) (Stuttgart, Germany).

HbA1c was measured by turbidimetric inhibition immunoassay (Roche Cobas c513 analyzer using the Tina quant® HbA1c Gen. 3 assay, Germany). MiniMed 780GTM data uploaded to CareLinkTM personal software during the follow-up by individuals who provided constent for their data to be aggregated were analyzed (CareLink; https://carelink.medtronic.eu). Time in range (TIR: 70-180 mg/dl), time below range (TBR: 70 mg/dl), time above range (TAR: >180 mg/dl), coefficient of variation (CV), glucose management indicator (GMI), sensor usage, time spent in AHCL and mean sensor glucose values were evaluated. Active insulin time was 2,5 hours and the target blood glucose value as 100 mg/dl in all patients at the initiation of AHCL and changed when necessary.

Statistical analyses were conducted using Statistical Package for the Social Sciences version 25.0 (SPSS Inc., Chicago, IL, USA). The level of significance was defined as p<0.05. Categorical variables were represented as counts and percentage values. Normal distribution was tested for quantitative variables. Continuous variables with normal or skewed distribution were presented as mean (standard deviation) or median (interquartile range). Group differences were investigated using the independent t-test for normally distributed data, the Mann-Whitney test for skewed data, and the chi-square tests used for categorical variables. Repeated values differences were investigated using One Way Anova for normally distributed data and the Friedman test for skewed data.

ELIGIBILITY:
Inclusion Criteria:

Use an advanced hybrid closed-loop system pump therapy (MiniMed 780G™, Medtronic, Northridge, CA USA)

Exclusion Criteria:

No with major medical problems as

* celiac disease,
* cystic fibrosis,
* psychiatric disorders
* communication difficulties

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents, and young adults with type 1 diabetes on an advanced hybrid closed-loop system pump therapy (MiniMed 780G™,Medtronic, Northridge, CA USA) ) receiving care at the Pediatric Endocrinology and Diabetes Clinic of Ege University (Izmir, Turkey)
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Macronutrient intake distribution | Day1
  At the beginning of the follow-up, the macronutrient distribution of the participant diets will be evaluated for compliance with national and international guidelines.
Macronutrient intake distribution | 3rd month
  In the third month of the follow-up, the compliance of the macronutrient distribution of the participant's diets with national and international guidelines and the change from the beginning of the follow-up will be evaluated.
Macronutrient intake distribution | 6th month
  In the 6th month of the follow-up, the compliance of the macronutrient distribution of the participant's diets with national and international guidelines and the change from the beginning of the follow-up will be evaluated.
HbA1c | Day 1
  As a metabolic control parameter of the beginning of follow-up period
HbA1c | 3rd month
  As a metabolic control parameter at the 3rd month of the follow-up and the change from the beginning of the follow-up will be evaluated.
HbA1c | 6th month
  As a metabolic control parameter at the 6th month of the follow-up and the change from the beginning of the follow-up will be evaluated.
Time in range (Time in range is the amount of time you spend in the target blood glucose range) | Day1
  As a metabolic control parameter of beginning of the follow-up period
Time in range(Time in range is the amount of time you spend in the target blood glucose range) | 3rd month
  As a metabolic control parameter at the 3rd month of the follow-up and the change from the beginning of the follow-up will be evaluated.
Time in range(Time in range is the amount of time you spend in the target blood glucose range) | 6th month
  As a metabolic control parameter at the 6th month of the follow-up and the change from the beginning of the follow-up will be evaluated.
Body mass index (kg/m2) | Day1
  As a follow-up weight related issues parameter
Body mass index(kg/m2) | 3rd month
  As a follow-up weight related issues parameter
Body mass index(kg/m2) | 6th month
  As a follow-up weight related issues parameter

CONTACTS AND LOCATIONS:
Overall Officials: Yelda Mansuroglu, Study Chair — ege university department of pediatrics; Günay Demir, MSc, Study Chair — ege university department of pediatrics; Hanife Balkı, Dr, Study Chair — ege university department of pediatrics; Samim Özen, Assoc Prof Dr, Study Chair — ege university department of pediatrics; Sukran Darcan, Prof Dr, Study Chair — ege university department of pediatrics; Damla Goksen, Prof Dr, Study Director — ege university department of pediatrics; yasemin Atik-Altinok, PhD, Principal Investigator — ege university department of pediatrics
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University, Medical Faculty, Division of Pediatric Endocrinology, Izmir, Bornova
  - Ege University Faculty of Medicine Department of Pediatrics, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atik-Altinok Y, Mansuroglu Y, Demir G, Balki HG, Ozen S, Darcan S, Goksen D. Does minimed 780GTM insulin pump system affect energy and nutrient intake?: long-term follow-up study. Eur J Clin Nutr. 2024 Jul;78(7):615-621. doi: 10.1038/s41430-024-01422-y. Epub 2024 Mar 8. PMID 38459160